CLINICAL TRIAL: NCT06407206
Title: Effects of Sub Occipital Muscle Inhibition Technique in Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC OMAIRAH AIEN
Record Dates: First submitted 2024-04-29; First posted 2024-05-09 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Mechanical Low Back Pain
Keywords: mechanical low back pain; sub occipital muscle inhibition; hamstring flexibility
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub occipital muscle inhibition technique along with conventional therapy (Experimental): Patient is in supine position Therapist sits near the head of the participant and places his hand below the head of the participant With the pads of hand therapist palpates the arch of atlas between the occipital protuberance and spinous process of axis and place the middle and ring finger over it by flexing the metacarpophalangeal joint in 90 degrees of flexion, base of skull will rest on hands Pressure is exerted in upward direction towards the therapist and is maintained for two minutes so that the muscle scan relax Participants are guided to keep their eyes close in order to avoid movement which affects the tone of sub occipital muscle
  Interventions: Other: Sub occipital muscle inhibition technique and conventional therapy
- conventional therapy (Other): Transcutaneous electrical nerve stimulation at lower back and hamstring muscles (pulse rate: 4Hertz, pulse duration: 150µs for 15mins) Hot pack ( 15mins),Ankle pumps (15 reps with 5 sec hold), Knee Range of motions (flexion and extension,10 reps),Quadriceps set (10 reps,5 sec hold),Vastus Medialis oblique (10 reps 5 sec hold),Gluteus sets (10 reps, 5 sec hold),Single knee to chest (10 reps with 10 sec hold) McKenzie exercises (10 reps with 10 sec hold and 10 sec rest),Stretching of calf and hamstring muscles (passive stretching,7 reps with 5 sec hold).
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Sub occipital muscle inhibition technique and conventional therapy — Patient is in supine position Therapist sits near the head of the participant and places his hand below the head of the participant With the pads of hand therapist palpates the arch of atlas between the occipital protuberance and spinous process of axis and place the middle and ring finger over it by flexing the metacarpophalangeal joint in 90 degrees of flexion, base of skull will rest on hands Pressure is exerted in upward direction towards the therapist and is maintained for two minutes so that the muscle scan relax Participants are guided to keep their eyes close in order to avoid movement which affects the tone of sub occipital muscle
  Arms: Sub occipital muscle inhibition technique along with conventional therapy
Other: conventional therapy — Transcutaneous electrical nerve stimulation at lower back and hamstring muscles (pulse rate: 4Hertz, pulse duration: 150µs for 15mins) Hot pack ( 15mins),Ankle pumps (15 reps with 5 sec hold), Knee Range of motions (flexion and extension,10 reps),Quadriceps set (10 reps,5 sec hold),Vastus Medialis oblique (10 reps 5 sec hold),Gluteus sets (10 reps, 5 sec hold),Single knee to chest (10 reps with 10 sec hold) McKenzie exercises (10 reps with 10 sec hold and 10 sec rest),Stretching of calf and hamstring muscles (passive stretching,7 reps with 5 sec hold).
  Arms: conventional therapy

SUMMARY:
The aim of study is to determine the effects of sub occipital muscle inhibition technique in mechanical low back pain, hamstring muscle flexibility, lumbar ranges and functional disability. This study will focus on either this technique have effects on reliving lumbar pain, improving flexibility of hamstring muscles and lumbar ranges or not.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common health condition, 70% of population of all ages is suffering from low back pain. Females have higher prevalence of low back pain than males. Individuals with low back pain experience muscle stiffness tension and pain in the back of body between the lower edge of 12th rib and the lower border of gluteal creases in the lumbo-sacral area (from L1-S1 vertebra) with a duration of more than three months. Low back pain can be mechanical in nature and is not associated with any other pathology .The primary etiological factors of mechanical low back pain is repetitive trauma and overuse.

Hamstring is a multi - joint muscle complex which consists of three muscles ( semitendinosus, semimembranosus and biceps femoris muscle) that covers the posterior thigh extending from ischial tuberosity to the medial and lateral aspects of the knee joint, performing flexion of knee and extension of hip joint. Hamstring muscle is prone to tightness, its flexibility have a vital role in maintaining the normal lumbar spine mechanics. Hamstring tightness is common among ages of 18-25 years with about 62% to 82% prevalence .Hamstring shortening during spinal flexion limits anterior pelvic tilting resulting in higher compressive loads on lumbar spine. It will place extreme pressure on lumbar extensors, involved in maintaining pelvic motion which will result in LBP .

Sub occipital muscle inhibition technique is a technique that results in relaxing the tense fascia and sub occipital muscles .It can be relaxed by applying pressure to sub occipital region while patient is lying in supine position. It is able to relax the fascia and results in increasing hamstring flexibility, which further results in reducing low back pain, increasing lumbar spine mobility and reducing functional limitations

ELIGIBILITY:
Inclusion Criteria:

* Chronic mechanical low back pain > 12 weeks
* Patients with hamstring tightness having popliteal angle more than 30 degrees.
* Negative sacroiliac distraction test to exclude sacroiliac joint pain

Exclusion Criteria:

* Acute severe low back pain
* Patients with hamstring injury
* Active tumor or infection
* Fractures of cervical and lumbar spine
* History of previous lumbar, hip and knee surgery
* Migraine
* Fever
* Sacroiliac joint dysfunction
* Cauda equine syndrome
* Patients having cognitive or mental retardation

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Active knee extension test: | two weeks
  Active knee extension test is performed for assessing the flexibility of hamstring muscles. The test is performed by positioning the participant in supine position, hip is placed at 90 degrees of flexion while opposite leg is stabilized in order to avoid hip flexion. The lumbar spine is in neutral position. The fulcrum of goniometer is placed over the lateral condyle of femur, proximal arm of goniometer is placed on the lateral surface of femur keeping the greater trochanter for reference and the distal arm is placed along the lateral surface of fibula with lateral malleolus keeping for reference. The participant is then asked to actively extend the knee till the point of pain or maximum tolerable stretch to hamstring muscle, measurements are then recorded from goniometer. its reliability with intra-class correlation coefficient (ICC) of 0.87 for dominant knee and 0.81 for non-dominant knee. .
Numeric Pain Rating Scale (NPRS): | two weeks
  The Numeric Pain Rating Scale (NPRS) is used to measure the subjective intensity of pain. The NPRS is an eleven-point scale ranging from 0 to 10. In which "0" is for no pain and "10" is for the most intense/worst pain, while the NPRS exhibited moderate reliability (ICC = 0.27-0.84)
Inclinometer for range of motion | two weeks
  An inclinometer is a commonly used device in physiotherapy to measure angles and the range of motion (ROM) of joints.it consists of a sensor which is sensitive to gravity and measures the angles, angle is then displayed on a digital display or a dial. The angle of the inclinometer will change as the joint moves. The maximum angle reached is the ROM of the joint. Inter-rater reliability of inclinometer is ICCs 0.71-0.87.
Oswestry disability index questionnaire (ODI): | two weeks
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researcher use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. Questionnaire examines the level of disability in 10 everyday activities of daily living which includes pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social interaction, travel, employment/ homemaking. Each item consists of 6 statements which are scored from 0-5, 0 indicating least disability and 5 indicates the greatest, total score is calculated as a percentage, with 0% indicating no disability and 100% indicating the highest level of disability. Test-retest reliability was consistently high across studies (mean ICC value of 0.937 ± 0.032).

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Dr. Ali Therapy clinic, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No